CLINICAL TRIAL: NCT04947319
Title: An Open-label Phase II Study to Investigate the Efficacy, Safety, and Pharmacokinetics of Tirabrutinib in Patients With Primary Central Nervous System Lymphoma (PCNSL)
Brief Title: Study of Tirabrutinib (ONO-4059) in Patients With Primary Central Nervous System Lymphoma (PROSPECT Study)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ONO-4059-09
Record Dates: First submitted 2021-06-16; First posted 2021-07-01 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Refractory Primary Central Nervous System Lymphoma; Primary CNS Lymphoma
Keywords: Bruton's Tyrosine Kinase Inhibitor, BTKi, tirabrutinib, ONO-4059, PROSPECT
MeSH Terms: interventions — tirabrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Tirabrutinib monotherapy in patients with relapsed or refractory PCNSL (Part A) (Experimental): Patients with relapsed or refractory PCNSL who meet eligibility criteria will be enrolled to receive tirabrutinib monotherapy.
  Interventions: Drug: Tirabrutinib
- Tirabrutinib + MTR in patients with newly diagnosed, treatment naïve PCNSL (Part B, Arm 1) (Experimental): Patients with newly diagnosed treatment naïve PCNSL who meet eligibility criteria will be enrolled to receive tirabrutinib + methotrexate/temozolomide/rituximab (MTR)
  Interventions: Drug: Tirabrutinib
- Tirabrutinib + R-MPV in patients with newly diagnosed, treatment naïve PCNSL (Part B, Arm 2) (Experimental): Patients with newly diagnosed treatment naïve PCNSL who meet eligibility criteria will be enrolled to receive tirabrutinib + rituximab/methotrexate/procarbazine/vincristine (R-MPV)
  Interventions: Drug: Tirabrutinib

INTERVENTIONS:
Drug: Tirabrutinib — Part A: Tirabrutinib 480 mg, taken orally, once a day on an empty stomach. Tirabrutinib treatment may be continued until disease progression or clinically unacceptable toxicity is observed.
  Other Names: ONO-4059
  Arms: Tirabrutinib monotherapy in patients with relapsed or refractory PCNSL (Part A)
Drug: Tirabrutinib — Part B, Arm 1 - Tirabrutinib 320 mg or 480 mg, taken orally, once a day on an empty stomach in combination with an MTR induction regimen. Tirabrutinib with MTR treatment will be continued for 4 induction cycles (28-day/cycle), or until disease progression or clinically unacceptable toxicity is observed.
  For patients not receiving consolidation treatment following induction, tirabrutinib 480 mg will be continued until disease progression, unacceptable toxicities are observed, or the Investigator decides to stop treatment.
  Other Names: ONO-4059
  Arms: Tirabrutinib + MTR in patients with newly diagnosed, treatment naïve PCNSL (Part B, Arm 1)
Drug: Tirabrutinib — Part B, Arm 2 - Tirabrutinib 320 mg or 480 mg, taken orally, once a day on an empty stomach in combination with an R-MPV induction regimen. Tirabrutinib with R-MPV treatment will be continued for 4 induction cycles (28-day/cycle), or until disease progression or clinically unacceptable toxicity is observed.
  For patients not receiving consolidation treatment following induction, tirabrutinib 480 mg will be continued until disease progression, unacceptable toxicities are observed, or the Investigator decides to stop treatment.
  Other Names: ONO-4059
  Arms: Tirabrutinib + R-MPV in patients with newly diagnosed, treatment naïve PCNSL (Part B, Arm 2)

SUMMARY:
This study will evaluate the efficacy, safety, and pharmacokinetics of tirabrutinib monotherapy in patients with relapsed or refractory PCNSL (Part A), and tirabrutinib in combination with one of two different high dose methotrexate based regimens (methotrexate/ temozolomide/rituximab or rituximab/methotrexate/procarbazine/ vincristine) as first line therapy in patients with newly diagnosed, treatment naïve PCNSL (Part B)

ELIGIBILITY:
Inclusion Criteria (Part A)

1. Written informed consent by the patient prior to screening
2. Patients aged ≥ 18 years on the day of consenting to the study
3. Pathologic diagnosis of PCNSL
4. Relapse or refractory PCNSL with at least one prior high dose methotrexate (HD-MTX) based therapy for PCNSL
5. Measurable brain lesion with a minimum diameter > 1.0 cm in gadolinium enhanced magnetic resonance imaging (MRI) performed within 14 days before starting tirabrutinib treatment
6. Eastern Cooperative Oncology Group performance score (ECOG PS) of 0, 1 or 2
7. Life expectancy of at least 3 months
8. Adequate bone marrow, renal, and hepatic function

Inclusion Criteria (Part B)

1. Written informed consent by the patient prior to screening
2. Patients aged ≥ 18 years on the day of consenting to the study
3. Pathologic diagnosis of PCNSL within the past 3 months
4. No prior anti-tumor treatments for PCNSL
5. Patients who, in the opinion of the Investigator, are suitable to receive treatment with a high dose methotrexate containing regimen
6. Measurable brain lesion with a minimum diameter > 1.0 cm in gadolinium enhanced MRI performed within 14 days before starting study treatment
7. ECOG PS of 0, 1 or 2
8. Life expectancy of at least 6 months
9. Adequate bone marrow, renal, and hepatic function

Exclusion Criteria (Part A)

1. Intraocular PCNSL with no brain lesion
2. Patient who is intolerant of contrast enhanced MRI due to allergic reactions to contrast agents
3. Patient with non-B cell PCNSL
4. Patient with systemic presence of lymphoma
5. Prior chemotherapy within 21 days, nitrosourea within 42 days, an antibody drug with anticancer activity (e.g., rituximab) within 28 days, prior radiotherapy within 14 days, prior major invasive surgery within 28 days, or allogeneic stem cell transplant within 6 months before starting tirabrutinib treatment
6. Prior BTK inhibitor treatment
7. Prior investigational drugs (including treatment in clinical research, unapproved combination products, and new dosage forms) within 28 days or 5 half-lives, whichever is shorter, before starting tirabrutinib treatment
8. Concomitant systemic corticosteroid on an ongoing basis within 14 days before starting tirabrutinib treatment, with the exception of the following:

   * Equivalent of up to 10 mg/day of prednisone for a disease other than PCNSL
   * Equivalent of up to 50 mg/day of prednisone (equal to 8 mg/day of dexamethasone) for patients with lesions of the brain or spinal cord or both
9. Patient who has received a CYP3A4 inducer or P-gp inducer within 14 days before starting tirabrutinib treatment
10. Concomitant warfarin, any other warfarin derivative anticoagulant, vitamin K antagonists, novel oral anticoagulants, or antiplatelet therapy on an ongoing basis within 7 days before starting tirabrutinib treatment
11. Active malignancy, other than PCNSL requiring systemic therapy
12. Poorly controlled comorbidity, severe heart, severe lung disease, clinically significant liver diseases that could affect protocol compliance or safety or efficacy assessments
13. Patient with bleeding diathesis
14. Patients with a history of moderate or severe hepatic impairment
15. QTcF > 480 milliseconds or requirement for ongoing treatment with concomitant medications that prolong the QT interval
16. Active infection, including a HIV, cytomegalovirus infection or SARS-CoV-2, or has had, within 28 days before starting tirabrutinib treatment, an infection (other than nail trichophytosis) that requires hospitalization or an intravenous antibiotic
17. Prior history of hypersensitivity or anaphylaxis to tirabrutinib
18. Prior history of Stevens Johnson Syndrome or Toxic Epidermal Necrolysis
19. Medical history of organ allografts
20. Tests positive for HIV-1 antibody and HIV-2 antibody, human T-lymphotropic virus 1 antibody, hepatitis B (HB) antigen, or hepatitis C virus (HCV) antibody. Tests positive for HBs antibody or hepatitis B virus core protein antibody and has a result of at least detectable in a hepatitis B virus deoxyribonucleic acid assay despite testing negative for HBs antigen.
21. Patient is unable to swallow tablets; has malabsorption, malabsorption syndrome, or a comorbidity that affects gastric function; has undergone complete resection of the stomach or small intestine; has ulcerative colitis or symptomatic inflammatory bowel disease; or has partial or complete intestinal obstruction.
22. Women who are pregnant or lactating
23. Patient is found incapable of giving consent due to dementia or another such condition
24. Patient is found to be otherwise ineligible for the study by the Investigator or sub-Investigator.

Exclusion Criteria (Part B)

1. Intraocular PCNSL with no brain lesion
2. Patients for whom the selected backbone regimen medications (i.e, methotrexate/temozolomide/rituximab for MTR and rituximab/methotrexate/procarbazine/vincristine for R-MPV) are contraindicated
3. Patients with a history of intolerable toxicity, hypersensitivity, anaphylaxis to the selected backbone regimen medications
4. Patient who is intolerant of contrast enhanced MRI due to allergic reactions to contrast agents
5. Patient with non-B cell PCNSL
6. Patient with systemic presence of lymphoma
7. Prior chemotherapy within 21 days, nitrosourea within 42 days, an antibody drug with anticancer activity (e.g., rituximab) within 28 days, prior radiotherapy within 14 days, prior major invasive surgery within 28 days, or allogeneic stem cell transplant within 6 months before starting tirabrutinib treatment
8. Prior BTK inhibitor treatment
9. Prior investigational drugs (including treatment in clinical research, unapproved combination products, and new dosage forms) within 28 days or 5 half-lives, whichever is shorter, before starting tirabrutinib treatment
10. Concomitant systemic corticosteroid on an ongoing basis within 14 days before starting tirabrutinib treatment, with the exception of the following:

    * Equivalent of up to 10 mg/day of prednisone for a disease other than PCNSL
    * Equivalent of up to 50 mg/day of prednisone (equal to 8 mg/day of dexamethasone) for patients with lesions of the brain or spinal cord or both
11. Patient who has received a CYP3A4 inducer or P-gp inducer within 14 days before starting tirabrutinib treatment
12. Concomitant warfarin, any other warfarin derivative anticoagulant, vitamin K antagonists, novel oral anticoagulants, or antiplatelet therapy on an ongoing basis within 7 days before starting tirabrutinib treatment
13. Active malignancy, other than PCNSL requiring systemic therapy
14. Poorly controlled comorbidity, severe heart, severe lung disease, clinically significant liver diseases that could affect protocol compliance or safety or efficacy assessments
15. Patient with bleeding diathesis
16. Patients with a history of moderate or severe hepatic impairment
17. QTcF > 480 milliseconds or requirement for ongoing treatment with concomitant medications that prolong the QT interval
18. Active infection, including a HIV, cytomegalovirus infection or SARS-CoV-2, or has had, within 28 days before starting tirabrutinib treatment, an infection (other than nail trichophytosis) that requires hospitalization or an intravenous antibiotic
19. Prior history of hypersensitivity or anaphylaxis to tirabrutinib
20. Prior history of Stevens Johnson Syndrome or Toxic Epidermal Necrolysis
21. Medical history of organ allografts
22. Tests positive for HIV-1 antibody and HIV-2 antibody, human T-lymphotropic virus 1 antibody, HBs antigen, or HCV antibody. Tests positive for HBs antibody or hepatitis B virus core protein antibody and has a result of at least detectable in a hepatitis B virus deoxyribonucleic acid assay despite testing negative for HBs antigen.
23. Patient is unable to swallow tablets; has malabsorption, malabsorption syndrome, or a comorbidity that affects gastric function; has undergone complete resection of the stomach or small intestine; has ulcerative colitis or symptomatic inflammatory bowel disease; or has partial or complete intestinal obstruction.
24. Women who are pregnant or lactating
25. Patient is found incapable of giving consent due to dementia or another such condition
26. Patient is found to be otherwise ineligible for the study by the Investigator or sub-Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2021-12-29 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) (Part A) | 1 year
  Overall response rate is defined as the proportion of patients with a best overall response of Complete response (CR), Complete response - unconfirmed (CRu), or (=partial response (PR) as determined by an independent review committee according to the International PCNSL Collaborative Group (IPCG) criteria.
Tirabrutinib dose estimate (Part B) | 1 month
  Estimate of tirabrutinib dose in combination with each backbone induction regimen (MTR and R-MPV) based upon treatment related AEs, SAEs, and toxicities observed during the initial cycle of induction therapy in the dose-ranging phase
Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) during induction (Part B) | 4 months
  Adverse events at each visit with the NCI CTCAE v5.0 used as a guide for the grading of severity.
Complete response rate (CRR) (Part B) | 4 months
  Complete response rate is defined as the proportion of patients with a best overall response of CR or CRu as determined by an independent review committee according to the IPCG criteria.

SECONDARY OUTCOMES:
Duration of response (DOR) (Part A and B) | 2 years
  Duration of response is defined as the time between the date of first response (CR, CRu, or PR) and the date of the first PD according to the IPCG criteria, or date of death due to any cause, whichever occurs first.
Time to response (TTR) (Part A and B) | 1 year
  Time to response is defined as the time between the date of first administration of tirabrutinib and the date of first response (CR, CRu, or PR) as determined by IRC according to the IPCG criteria.
Best overall response (BOR) (Part A and B) | 1 year
  Best overall response based on independent review committee (IRC) response determination is defined as the best response and is derived programmatically based upon the visit responses determined by IRC from the date of administration of tirabrutinib to the date of PD as determined by IRC or the date of initiation of subsequent anticancer therapy for PCNSL, whichever occurs first.
Change in corticosteroid dose (Part A) | 2 years
  Descriptive statistics will be calculated for the actual corticosteroid dose and the change from baseline at each assessment point.
Incidence and severity of AEs and SAEs (Part A and B) | 2 years
  Adverse events at each visit with the NCI CTCAE v5.0 used as a guide for the grading of severity.
Laboratory abnormality profile of tirabrutinib as measured by incidence and severity of clinical laboratory abnormalities (Part A and B) | 2 years
  Results of laboratory tests
ECG parameters by 12 lead ECG (Part A and B) | 2 years
  Heart rate, RR and QT intervals, QTc (QTcF, QTcB), PR interval, and QRS width.
PK parameters (Cmax) of tirabrutinib in the plasma (Part A and B) | 29 days
PK parameters (Tmax) of tirabrutinib in the plasma (Part A and B) | 29 days
PK parameters (AUC) of tirabrutinib in the plasma (Part A and B) | 29 days

CONTACTS AND LOCATIONS:
Overall Officials: Project Leader, Study Director — Ono Pharmaceutical Co. Ltd
Locations (39):
- United States (39):
  - University of Alabama at Birmingham School of Medicine, Birmingham, Alabama
  - Mayo Clinic- Phoenix, Phoenix, Arizona
  - City of Hope Comprehensive Breast Cancer Center, Duarte, California
  - University of California, Irvine, Irvine, California
  - Stanford University, Palo Alto, California
  - University of Colorado Denver, Aurora, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Georgetown University, Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - Mayo Clinic- Jacksonville, Jacksonville, Florida
  - University of Miami-Sylvester Cancer Center, Miami, Florida
  - Orlando Health, Orlando, Florida
  - Moffitt Cancer Center- Miami, Pembroke Pines, Florida
  - Piedmont Healthcare, Atlanta, Georgia
  - University of Kentucky, Lexington, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute - Brigham & Women's Hospital, Boston, Massachusetts
  - University Of Michigan, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - The University of Kansas Cancer Center (KUCC) (Kansas City Cancer Center (KCCC)) - North, Kansas City, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hackensack University Medical Center - John Theurer Cancer, Hackensack, New Jersey
  - Roswell Park Comprehensive Cancer Center (RPCCC) (Roswell Park Cancer Institute (RPCI)), Buffalo, New York
  - Memorial Sloan Kettering, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - Levine Cancer Center, Charlotte, North Carolina
  - Duke University School of Medicine, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Providence Health Cancer Center, Portland, Oregon
  - Penn State Hershey Cancer Center, Hershey, Pennsylvania
  - Abramson Cancer Center University of Pennsylvania, Philadelphia, Pennsylvania
  - Hillman Cancer Center, University of Pittsburgh, Pittsburgh, Pennsylvania
  - Lifespan Rhode Island Hospital, Providence, Rhode Island
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Houston Methodist Research Institute (HMRI), Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - The University of Utah - Huntsman Cancer Institute (HCI), Salt Lake City, Utah
  - The University of Vermont - Fletcher Allen Health Care, Burlington, Vermont
  - Seattle Cancer Care Alliance, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor maintained study web address — https://www.theprospectstudy.com/